CLINICAL TRIAL: NCT00042146
Title: Behavioral and Pharmacological Treatment for Insomnia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH060413 (NIH); R01MH060413 (NIH); DATR A4-GPS; NCT00218738 (obsolete NCT alias)
Record Dates: First submitted 2002-07-24; First posted 2002-07-26 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: Insomnia; Sleep Disorders; Sleep Deprivation
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders; Sleep Deprivation | interventions — Cognitive Behavioral Therapy; Zolpidem

INTERVENTIONS:
Behavioral: Cognitive-behavior therapy
Drug: zolpidem

SUMMARY:
This study will evaluate the long- and short-term effects of cognitive-behavior therapy (CBT), alone and in combination with zolpidem (Ambien®), for chronic insomnia.

DETAILED DESCRIPTION:
Insomnia is a prevalent health concern which is often associated with functional impairments, reduced quality of life, and increased health-care costs. The proposed study may provide useful information about optimal models for integrating behavioral and pharmacological therapies for the clinical management of insomnia.

Participants are randomly assigned to CBT or CBT plus medication. After the 6-week acute treatment phase, participants enter into a 6-month extended treatment phase. Of those treated with CBT alone initially, responders are randomized to extended CBT or no treatment. Of those receiving the combined CBT plus medication approach initially, responders are randomized to an extended treatment consisting of either CBT plus medication (used on an as needed schedule) or CBT alone (plus medication tapering). Outcome is evaluated across measures of sleep, clinical ratings, and several indices of daytime functioning. The measures are administered at baseline, at the end of the acute and extended treatment phases, and at 6, 12, and 24-month follow-up.

ELIGIBILITY:
Inclusion criteria:

* Subjective complaint of difficulties initiating or maintaining sleep, accompanied by marked distress or daytime impairments due to insomnia
* Sleep difficulties present 3 nights or more per week and lasting for more than 6 months

Exclusion criteria:

* Major medical or psychiatric problems

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2001-12

CONTACTS AND LOCATIONS:
Locations (1):
- Laval University, Québec, Quebec, Canada

REFERENCES:
- [Derived] Rochefort A, Jarrin DC, Belanger L, Ivers H, Morin CM. Insomnia treatment response as a function of objectively measured sleep duration. Sleep Med. 2019 Apr;56:135-144. doi: 10.1016/j.sleep.2019.01.016. Epub 2019 Jan 31. PMID 30871960
- [Derived] Beaulieu-Bonneau S, Ivers H, Guay B, Morin CM. Long-Term Maintenance of Therapeutic Gains Associated With Cognitive-Behavioral Therapy for Insomnia Delivered Alone or Combined With Zolpidem. Sleep. 2017 Mar 1;40(3):zsx002. doi: 10.1093/sleep/zsx002. PMID 28364426
- [Derived] Morin CM, Beaulieu-Bonneau S, Belanger L, Ivers H, Sanchez Ortuno M, Vallieres A, Savard J, Guay B, Merette C. Cognitive-behavior therapy singly and combined with medication for persistent insomnia: Impact on psychological and daytime functioning. Behav Res Ther. 2016 Dec;87:109-116. doi: 10.1016/j.brat.2016.09.002. Epub 2016 Sep 13. PMID 27658218
- [Derived] Morin CM, Vallieres A, Guay B, Ivers H, Savard J, Merette C, Bastien C, Baillargeon L. Cognitive behavioral therapy, singly and combined with medication, for persistent insomnia: a randomized controlled trial. JAMA. 2009 May 20;301(19):2005-15. doi: 10.1001/jama.2009.682. PMID 19454639